CLINICAL TRIAL: NCT04282577
Title: Urinary Nephrin and Alpha One Microglobulin as Early Renal Injury Biomarkers in Patients With Inflammatory Bowel Disease
Brief Title: Urinary Biomarkers of Renal Injury in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Gamal Abdelmalik, assistant lecturer, Assiut University
Other Study IDs: Kidney in IBD
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with chron's disease
  Interventions: Diagnostic Test: urinary nephrin and alpha one microglobulin
- patients with ulcerative cholitis
  Interventions: Diagnostic Test: urinary nephrin and alpha one microglobulin

INTERVENTIONS:
Diagnostic Test: urinary nephrin and alpha one microglobulin — urinary nephrin and alpha one microglobulin are biomarkers of glomerular filtration barrier injury and tubular injury respectively measured by ELISA

SUMMARY:
The study aims to early detection of renal injury in patients diagnosed to have inflammatory bowel disease with normal kidney function test focusing on glomerular filtration barrier injury and tubular injury and it's relation to disease activity so precautions could be taken properly to prevent further renal injury later on .

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic and relapsing inflammatory condition of the gastrointestinal tract. Crohn's disease and ulcerative colitis are the two principal types of IBD. The prevalence of IBD has been increasing worldwide . Extraintestinal manifestations of IBD are common, occurring in 6% to 47% of patients involving nearly every organ system .

Renal and urinary system involvement are common in IBD patients with incidence varying from 4% to 23% and is greater in patients with more severe and long-standing disease. Apart from secondary complications, such as nephrolithiasis, hydronephrosis and amyloidosis, other disorders have also been reported. Membranous glomerulonephritis, rapidly progressive glomerulonephritis, mesangiocapillary glomerulonephritis, IgA nephropathy, thin basement membrane disease and kidney granuloma found to be connected with IBD. In addition, non-specific morphological changes in the glomeruli of patients with IBD, like podocyte effacement and mesangial deposition of immunoglobulin and complement have been well documented. Cases of interstitial nephritis reported to be attributed to the nephrotoxic effect of aminosalicylates which used in IBD treatment.

Alpha one microglobulin is a relatively small protein that undergoes glomerular filtration followed by reabsorption and catabolism in the proximal tubules. Increased urinary α1-microglobulin concentration therefore provides an index of proximal tubule dysfunction .

Glomerular filtration barrier related protein changes have not been closely investigated in IBD patients . Nephrin is podocyte-associated protein that play key roles in maintaining the structural and functional integrity of the kidney's filtration barrier. The shedding of nephrin reflects compromisation of podocytes' functional and structural integrity.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed to have inflammatory bowel disease (ulcerative colitis or chron's disease )with age more than 18 years and normal kidney function test

Exclusion Criteria:

Patients known to have renal disease due to other causes . Diabetic patients . Hypertensive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inflammatory bowel disease patients aging more than 18 with no concomitent kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Early detection of renal injury in patients diagnosed to have inflammatory bowel disease with normal kidney function | baseline
  using urinary biomarkers (nephrin and alpha one microglobulin ) for early detection of renal injury in inflammatory bowel disease patients

REFERENCES:
- [Background] Akankwasa G, Jianhua L, Guixue C, Changjuan A, Xiaosong Q. Urine markers of podocyte dysfunction: a review of podocalyxin and nephrin in selected glomerular diseases. Biomark Med. 2018 Aug;12(8):927-935. doi: 10.2217/bmm-2018-0152. Epub 2018 Jul 6. PMID 29976076
- [Background] Chang CJ, Wang PC, Huang TC, Taniguchi A. Change in Renal Glomerular Collagens and Glomerular Filtration Barrier-Related Proteins in a Dextran Sulfate Sodium-Induced Colitis Mouse Model. Int J Mol Sci. 2019 Mar 22;20(6):1458. doi: 10.3390/ijms20061458. PMID 30909435